CLINICAL TRIAL: NCT04445636
Title: Efficacy of Dexmedetomidine Versus Morphine as an Adjunct to Bupivacaine in Caudal Anesthesia for Pediatric Thoracic Surgeries. A Randomized Controlled Trial.
Brief Title: Efficacy of Dexmedetomidine Versus Morphine as an Adjunct to Bupivacaine in Caudal Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelaziz Ismail, Director, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N239-2020
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia, Local
Keywords: thoracic surgeries; pediatric caudal; dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be achieved by a statistician using an online random number generator. Patient codes will be placed into sequentially numbered sealed opaque envelopes by a research assistant who is not involved in the study. An anesthesia resident not involved in patient management will be responsible for opening the envelope. The anesthesia resident will prepare the study drug according to the instructions contained within each envelope and give it to the anesthesiologist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): A group which will receive dexamedetomidine as an adjunct to bupivacaine used in caudal anesthesia.
  Interventions: Drug: Dexmedetomidine
- Morphine group (Experimental): A group which will receive morphine as an adjunct to bupivacaine used in caudal anesthesia.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Dexmedetomidine — Caudal block with Dexametomedine as an adjuvant to bupivacaine.
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Morphine — Addition of morphine as adjuvant to bupivacaine during caudal block.
  Arms: Morphine group

SUMMARY:
The aim of this study is to compare the duration of postoperative analgesia, and any side effects of caudal dexmedetomidine versus morphine in combination with bupivacaine in pediatric patients undergoing thoracic surgeries.

DETAILED DESCRIPTION:
The patients will be randomized in a blinded fashion to get enrolled into 2 equal groups: Group A patients (n =25) will receive caudal epidural analgesia using dexmedetomidine with bupivacaine, whereas Group B patients (n = 25) will receive caudal epidural analgesia using morphine with bupivacaine.

Randomization will be achieved by using an online random number generator. Patient codes will be placed into sequentially numbered sealed opaque envelopes by a research assistant who is not involved in the study. An anesthesia resident not involved in patient management will be responsible for opening the envelope. The anesthesia resident will prepare the study drug according to the instructions contained within each envelope and give it to the anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II, III.
* Patients undergoing lung cyst excision.
* Patients undergoing Patent Ductus Arteriosus ligation.

Exclusion Criteria:

* Preoperative mechanical ventilation.
* Preoperative inotropic support
* History of mental retardation or delayed development that may interfere with pain intensity assessment
* Known or suspected coagulopathy,
* Any congenital anomalies of the sacrum or any infection at the site of injection.
* Known or suspected allergy to any of the studied drugs.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia in hours. | 3 months
  Duration of postoperative analgesia in hours.

SECONDARY OUTCOMES:
Opioid consumption in the first 24 hours post- operative. | 3 months
  Opioid consumption in the first 24 hours post- operative.
The duration of ICU stay in days | 3 months
  The duration of ICU stay in days
Pain score FLACC from 0 to 6 | 3 months
  Pain score FLACC from 0 to 6
Post operative heart rate | 3 months
  Postoperative heart rate in beat per minute

CONTACTS AND LOCATIONS:
Overall Officials: AHMED ISMAIL, Lecturer, Study Director — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The patients data are confidential

REFERENCES:
- [Background] Anand VG, Kannan M, Thavamani A, Bridgit MJ. Effects of dexmedetomidine added to caudal ropivacaine in paediatric lower abdominal surgeries. Indian J Anaesth. 2011 Jul;55(4):340-6. doi: 10.4103/0019-5049.84835. PMID 22013248
- [Background] El Shamaa HA, Ibrahim M. A comparative study of the effect of caudal dexmedetomidine versus morphine added to bupivacaine in pediatric infra-umbilical surgery. Saudi J Anaesth. 2014 Apr;8(2):155-60. doi: 10.4103/1658-354X.130677. PMID 24843324
- [Background] Nguyen KN, Byrd HS, Tan JM. Caudal analgesia and cardiothoracic surgery: a look at postoperative pain scores in a pediatric population. Paediatr Anaesth. 2016 Nov;26(11):1060-1063. doi: 10.1111/pan.12990. Epub 2016 Aug 23. PMID 27550555